CLINICAL TRIAL: NCT02382328
Title: Effectiveness of Alpha Lipoic Acid on Clinical and Electrophysiological Recovery in Patients With Carpal Tunnel Syndrome Surgical Release
Brief Title: Alpha Lipoic Acid on Clinical and Electrophysiological Recovery in Carpal Tunnel Syndrome Undergoing Surgical Release
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Elisa Alejandra Monroy Guizar, Medico Especialista Medicina de Rehabilitación, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 265/14
Record Dates: First submitted 2015-02-18; First posted 2015-03-06 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- alpha lipoic acid (Experimental): 600mg/24 oral pills alpha lipoic acid 28 days before and 120 days after carpal tunnel release.
  Interventions: Drug: alpha lipoic acid
- Placebo (Placebo Comparator): Oral pills of mangensium inactivated 28 days before and 120 days after carpal tunnel release.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: alpha lipoic acid — comparison of 600mg/24h oral, alpha lipoid acid, 28 days before and 120 days after surgery (carpal tunnel release) versus placebo in carpal tunnel syndrome patients.
  Other Names: thiocitic acid
  Arms: alpha lipoic acid
Drug: Placebo — Placebo oral pills, 28 days before and 120 days after surgery (carpal tunnel release) versus placebo in carpal tunnel syndrome patients.
  Other Names: inactive magnesium
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the effectiveness of use Alpha lipoic acid before and after surgical release of carpal tunnel syndrome. Controlled Clinical trial.

DETAILED DESCRIPTION:
The main purpose of this study is to determine the effectiveness of using an oral supplementation of alpha lipoid acid to improve clinical and electrophysiological recovery after carpal tunnel release surgery. This research is designed as a double blinded clinical trial, with a calculated sample size of 40 patients, divided in two groups of 20 (A placebo, B alpha lipoid acid). All patients will undergo open carpal tunnel release surgery, the procedure will be performed by an expert surgeon. A total of four visits will be performed as follows: T0. baseline 4 weeks before surgery, T1 immediately before surgery, T2: 4 weeks after surgery, T3: 8 weeks after surgery, T4: 12 weeks after surgery. The assessment to be perform on each visit includes: physical examination, Boston Questionary for Carpal Tunnel Syndrome. Nerve conduction study and ecographic evaluation will be performed on visits T0, T1 and T4. Statistical Analysis: Categorical variables will be assessed as counts and percent frequency and compared using the chi-squared test. All statistical analyses will be performed using the SPSS 21.0 package (SPSS Inc., Chicago, IL, USA). A two-tailed P value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* clinical and electrophysiological diagnosis of carpal tunnel syndrome

Exclusion Criteria:

* rheumatic diseases
* distal radio or carpal fractures.
* pregnant women
* alpha lipoid acid allergy
* local injections (ej. steroid carpal injections)
* peripheral nervous system diseases (which may cause nerve conduction study abnormalities).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
median nerve sensory latency (using nerve conduction studies to determine median sensory latency.) | 120 days after surgery
  using nerve conduction studies to determine median sensory latency.

SECONDARY OUTCOMES:
cross sectional area of median nerve (sonographic measurement to determine cross sectional area of median nerve.) | 120 days after surgery
  sonographic measurement to determine cross sectional area of median nerve.

CONTACTS AND LOCATIONS:
Overall Officials: Leonel Garcia, PhD, Study Director — University of Guadalajara
Locations (1):
- Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Pajardi G, Bortot P, Ponti V, Novelli C. Clinical usefulness of oral supplementation with alpha-lipoic Acid, curcumin phytosome, and B-group vitamins in patients with carpal tunnel syndrome undergoing surgical treatment. Evid Based Complement Alternat Med. 2014;2014:891310. doi: 10.1155/2014/891310. Epub 2014 Jan 19. PMID 24563654
- [Result] Di Geronimo G, Caccese AF, Caruso L, Soldati A, Passaretti U. Treatment of carpal tunnel syndrome with alpha-lipoic acid. Eur Rev Med Pharmacol Sci. 2009 Mar-Apr;13(2):133-9. PMID 19499849